CLINICAL TRIAL: NCT06469827
Title: Evaluation of Consciousness Impairment in Severe TBI and Full-cycle Neuroregulation Based on Multimodal Imaging
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Ankang Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-567
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury
Keywords: severe traumatic brain injury; multimodal imaging; brain injury recovery; neuroregulation; disorder of consciousness
MeSH Terms: conditions — Brain Injuries, Traumatic; Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about in Evaluation of consciousness impairment in severe TBI and full-cycle neuroregulation based on multimodal imaging. The main question it aims to answer is:

•For the existing examination means of super early neurological consciousness level recognition and function assessment accuracy of poor technical bottleneck, different period individual target brain space positioning difficulties and single rehabilitation technology of whole cycle rehabilitation system, with severe TBI patients as the research object.

DETAILED DESCRIPTION:
Brain trauma (traumatic brain injury, TBI) is one of the most common acute and severe diseases in neurosurgery. It has the characteristics of high disability rate and high mortality rate, and has become a major global medical and public health problem. Disorder of consciousness (Disorder of consciousness, DOC) is one of the most common clinical manifestations in the early stage of severe TBI patients with coma. Long-term DOC is the main manifestation of poor prognosis and can cause disability or death. Up to 43% of patients diagnosed with vegetative patients were reclassified as minimal consciousness. How to realize the accurate assessment of DOC population consciousness state, strengthen the early identification and functional assessment of people with severe TBI, and establish the whole-process rehabilitation system and management strategy for severe neurological diseases are the main clinical concerns. This project for the existing examination means of super early neurological consciousness level recognition and function assessment accuracy of poor technical bottleneck, different period individual target brain space positioning difficulties and single rehabilitation technology of whole cycle rehabilitation system, with severe TBI patients as the research object.

The specific research was mainly conducted from the following three aspects: (1) the relationship between EEG qualitative power spectrum typing, quantitative power spectrum index and behavioral scale, and the assessment of early awareness recovery in DOC patients; (2) the auxiliary scheme for ICU based on near-infrared light therapy; (3) the light-magnetic combined neuroregulation strategy for subacute patients based on precise positioning of fMRI in the resting state.

ELIGIBILITY:
Inclusion Criteria:

1. GCS 3-8 points
2. Loss of consciousness greater than 6 hours or consciousness and coma greater than 6 hours within 24 hours after injury

Exclusion Criteria:

1. Alcohol consumption, substance abuse during or within the previous 24 hours
2. Previous history of traumatic brain injury, MRI contraindication, penetrating brain injury, psychotropic substance use, spinal cord injury, positive neurological examination, multifunctional disorder
3. Previous history of traumatic brain injury, MRI contraindication, penetrating brain injury, psychotropic substance use, spinal cord injury, positive neurological examination, multifunctional disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population was in patients over 18 years of age with severe TBI. Inclusion Criteria: 1. GCS 3-8 points. 2. Loss of consciousness greater than 6 hours or consciousness and coma greater than 6 hours within 24 hours after injury. Exclusion Criteria: 1. Alcohol consumption, substance abuse during or within the previous 24 hours. 2. Previous history of traumatic brain injury, MRI contraindication, penetrating brain injury, psychotropic substance use, spinal cord injury, positive neurological examination, multifunctional disorder.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Full Outline of Unresponsiveness, FOUR | At 0,2,4,6,8, and 10 days after treatment
  The FOUR is an questionnaire which has four main assessments: eye opening, exercise, brain stem reflex, and respiratory function. Each item has a full score of 4 and a total score of 16. Brainstem reflex and respiratory function of FOUR are more sensitive than the GCS language score for predicting mortality risk in ICU patients. The total score was 0 to 16, with lower scores indicating a greater probability of death and disability.
Sensory Modality Assessment and Rehabilitation Technique, SMART | At 0,2,4,6,8, and 10 days after treatment
  Assessment of sensory patterns (Sensory Pattern Assessment) and rehabilitation techniques are commonly used in rehabilitation therapy to assess the sensory function and motor ability of patients to develop personalized rehabilitation programs.
  Sensory pattern assessment usually involves the following steps:
  1. Assess the patient's sensory function.
  2. Evaluation sensory conduction pathways.
  3. Evaluation of sensory patterns.
  Assessment of rehabilitation techniques usually involves the following steps:
  1. Assess the patient's motor function.
  2. Evaluation of exercise mode.
  3. Develop rehabilitation plan.
Coma Recovery Scale Revised, CRS-R | At 0,2,4,6,8, and 10 days after treatment
  The CRS-R score is a clinical tool used to assess the level of consciousness in comatose and drowsy patients, fully called the Coma Recovery Scale-Revised. The scoring tool includes 23 items covering different aspects of the patient, such as vision, hearing, motor, response, etc. By scoring these items, medical professionals can assess patient level of awareness and response capacity in order to develop corresponding treatment and rehabilitation plans.
  Auditory function scale = for movement to commands. 4-Consistent Movement to Command 3-Reproducible Movement to Command 2-Localization to Sound
  1-Auditory Startle 0-None

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No